CLINICAL TRIAL: NCT05499793
Title: Impact of Zingiber Officinale on Symptoms and Hormonal Changes During the Menopausal Period in Duhok -Iraq
Brief Title: Impact of Ginger on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Niroosh Hashim Taha, MSc Student in clinical Pharmacology, University of Duhok
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24102021-10-36
Record Dates: First submitted 2022-08-07; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Menopause
MeSH Terms: interventions — ginger extract

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: A pharmacist professional was responsible for distributing the treatment (ginger) and placebo and he was in charge to assign the participants to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Ginger) (Experimental): All the participants were given Zingiber Officinale powder (500 mg) capsules twice daily for twelve weeks.
  Zingiber Officinale capsules were purchased from Pure Mountain Botanicals, 1712 Pioneer Ave # 1139 Cheyenne Wyoming 82001 (USA)
  Interventions: Dietary Supplement: Zingiber Officinale powder
- Control group (Placebo) (Placebo Comparator): All the participants were given starch powder (50 mg) capsules twice daily for twelve weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zingiber Officinale powder — Ginger powder
  Other Names: Ginger
  Arms: Treatment group (Ginger)
Dietary Supplement: Placebo — Starch powder
  Other Names: control
  Arms: Control group (Placebo)

SUMMARY:
This study aimed to examine the impact of one gram of Zingiber Officinale powder on menopausal symptoms since a large number of menopausal women in this region (Duhok city in the North of Iraq) are reluctant to take the conventional treatment for improving their menopausal symptoms and they prefer of taking the ginger powder and surprisingly many of those patients reported positive effects on their symptoms and general well being.

DETAILED DESCRIPTION:
After taking the scientific and ethical approval from the College of the Pharmacy/ University of Duhok and the Directorate of Duhok Health (reference number 24102021-10-36) to look at the impact of Zingiber officinale on menopausal symptoms in women between 45 and 60 years old. A clinical interventional study was launched at the Gynecology Department in Azadi Teaching Hospital in Duhok Governorate, Iraq, from December 2021 to May 2022. This study initially recruited seventy women who matched the inclusion criteria. All the recruited women were informed about the study protocols, and they had the option to withdraw from it anytime. After giving written consent, they were randomly divided into one of two research groups through a random number generator software. Thirty-five women functioned as controls and were given placebo capsules for twelve weeks (A professional pharmacist formulated a 50mg starch purchased from the local market to look similar to the ginger capsule). The other thirty-five women were given pure Zingiber Officinale powder (500mg) in capsules twice daily for twelve weeks (Zingiber Officinale capsules were purchased from Pure Mountain Botanicals, 1712 Pioneer Ave # 1139 Cheyenne Wyoming 82001 (USA)). Twenty women completed the study in the placebo group, while thirty women completed the survey in the Ginger group. Unfortunately, fifteen participants from the control group and five women from the treatment group didn't finish the study and were excluded as they were not tighter to the project protocol.

The frequency and severity of menopausal symptoms were assessed using an internationally recognized questionnaire menopausal rating scale (MRS). Percentage differences between pre-treatment were compared to post-treatments.

The serum estrogen, progesterone, FSH, and LH levels were measured before and after treatment using a suitable kit for each hormone by Cobas e 411 analyzers (Roche Diagnostics).

ELIGIBILITY:
Inclusion Criteria:

* Women living in Duhok city with self-reported menopause symptoms
* Aged between 45 and 60 years

Exclusion Criteria:

* Not on treatment for menopausal symptoms
* Patients Having chronic diseases like hypertension, Ischemic heart diseases or Diabetes mellitus
* Patients having coagulopathies
* Patient's having hormone-dependent malignancies

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Impact of Zingiber Officinale on hot flush in menopausal women | six weeks treatment with Zingiber Officinale powder
  A significant change in the intensity of hot flushes was observed in the menopausal rating scale in menopausal women treated with ginger powder compared to pre-treatment.
Impact of Zingiber Officinale on Night sweating in menopausal women | six weeks treatment with Zingiber Officinale powder
  A significant change in the intensity of night sweating was observed in the menopausal rating scale in menopausal women treated with ginger powder compared to pre-treatment.
Impact of Zingiber Officinale on estrogen levels in menopausal women | six weeks treatment with Zingiber Officinale powder
  A significant change was observed in serum estrogen levels in menopausal women treated with ginger powder compared to pre-treatment.
Impact of Zingiber Officinale on body weight in menopausal symptoms | six weeks treatment with Zingiber Officinale powder
  A significant change was observed in body weight in kilograms in menopausal women treated with ginger powder compared to pre-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Duhok College of Pharmacy, Duhok, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
The collected Data will not be shared until the study has been published